CLINICAL TRIAL: NCT04218955
Title: Parental Acceptance and Perception of Silver Diamine Flouride Application Among A Sample of Egyptian Children
Brief Title: Parental Acceptance and Perception of Silver Diamine FlouridApplication Among A Sample of Egyptian Children.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Abd El Aziz Waly, Dentist, Cairo University
Other Study IDs: Parental acceptance of SDF
Record Dates: First submitted 2019-12-27; First posted 2020-01-06 (Actual); Last update posted 2020-01-06 (Actual); Status verified 2019-12

CONDITIONS: Early Childhood Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Asking parents if they can accept staining from treat their children by silver Diamine Flouride or Not
  Interventions: Combination Product: Silver Diamine Flouride

INTERVENTIONS:
Combination Product: Silver Diamine Flouride — Material used to arrest caries in children

SUMMARY:
Dental caries can be prevented or arrested . Moreover, preventive measures for dental caries are more cost effective than emergency room visits or restorative treatments when the illness has been established . One of the recent preventive methods of dental caries is silver diamine flouride . SDF has been used as an alternative treatment for caries prevention and arrest . Several studies showed that silver diamine flouride cause staining of the treated teeth . However, parents have different attitudes toward using SDF considering its positives and negatives.

DETAILED DESCRIPTION:
Dental caries is one of the most common diseases in the world, with a prevalence of 69%-79% . Early childhood caries (ECC) has been recognized by the American Dental Association as an important public health issue and was defined as presence of 1 or more decayed, missing, or filled tooth surfaces (dmfs) in any primary tooth in a preschool-aged child . Caries was known to be managed through two main approaches: Treatment, which includes drill and fill which is a challenge specially in minimally cooperative children and the second approach is prevention which depends on cease the process of caries formation at an early stage which is more effective . One of the recently marketed preventive measures of dental caries is silver diamine fluoride (SDF) .

In 2014, SDF was approved by the US Food and Drug Administration as a treatment for dentinal sensitivity .It was proven to be a cost-effective, minimally invasive, and handy treatment . Silver diamine flouride is easy to apply in a minimally cooperative individual . More important, it has shown a noticeable success rate in caries prevention, especially in early childhood caries cases . It provides families with an alternative solutions for managing dental caries, particularly if caries was detected at an early stage . Moreover, it could save time and effort for both families and dental teams.

The major downside of SDF is the unesthetic permanent black discoloration of the arrested lesion , which could affect parental acceptance for the treatment and may result in shifting to another esthetically acceptable treatment.

ELIGIBILITY:
Inclusion Criteria:

* parents whose children with early childhood caries. Accepting participations.

Exclusion Criteria:

* Refusal of participation.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Parents whose children have early childhood caries seeking for dental treatment coming to the outpatient diagnostic clinics in the department of pediatric dentistry, Cairo University, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-03-01 (Estimated)

PRIMARY OUTCOMES:
Parental Satisfication about treat their children with silver Diamine flouride | Baseline
  Using Likert scale ranging from Strong Accept ,Accept ,Neutral, Refuse, Strong Refuse.